CLINICAL TRIAL: NCT06678555
Title: A Retrospective Study to Evaluate the Real-World Effectiveness of Lorlatinib Among ROS1-Positive NSCLC Patients
Brief Title: A Study to Learn About Lorlatinib in Patients With Non-Small Cell Lung Cancer (NSCLC) Which Has Spread Out.
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B7461048; NCT06678555 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — lorlatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lorlatinib: Patients with ROS1(+) advanced/metastatic NSCLC had been treated with lorlatinib.
  Interventions: Drug: Lorlatinib

INTERVENTIONS:
Drug: Lorlatinib — Lorlatinib is an ALK/ROS1 tyrosin kinase inhibitor.
  Other Names: PF-6463992

SUMMARY:
The purpose of this study is to learn about lorlatinib for the possible treatment of lung cancer which could not be controlled.

This study is seeking participants who:

* have lung cancer that could not be controlled.
* have a type of gene called a ROS proto-oncogene 1. A gene is a part of your DNA that has instructions for making things your body needs to work.
* have received at least 1 treatment before.

All participants in this study had received lorlatinib. Lorlatinib is a tablet that is taken by mouth at home. They continued to take lorlatinib until their cancer was no longer responding. The study will look at the experiences of people receiving the study medicine. This will help to see if the study medicine is safe and effective.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are aged 18 years or older on index date
2. Patients have confirmed diagnosis of ROS1-positive NSCLC
3. Patients have received at least one dose of lorlatinib between 1st April, 2018, and 30th September, 2023

Exclusion Criteria:

1. Patients participated in any clinical trials using lorlatinib during the observation period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective, observational study to investigate effectiveness, treatment patterns, and gene mutation profile of ROS1-positive NSCLC patients who had received lorlatinib after any TKI treatment failure in Taiwan using an EMR database, NTUH-iMD. Study population consists of patients who were diagnosed with ROS1-positive NSCLC and received at least one dose of lorlatinib between 1st April, 2018, and 30th September, 2023 after any TKI treatment failure.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2025-07-04 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
real-world progression-free survival | 74 months from 1st April, 2018
  Time to real-world disease progression or death, whichever occurs first, during observation period from index date will be summarized by the K-M plot with the corresponding 95% CI.
  Index date is the date of the first dose of lorlatinib.
The overall survival (OS) | 74 months from 1st April, 2018
  Time to death during observation period from index date will be summarized by the K-M plot with the corresponding 95% CI.
  Index date is the date of the first dose of lorlatinib.
The real world time to next treatment (rwTTNT) | 74 months from 1st April, 2018
  Time to subsequent treatment or death, whichever occurs first, during observation period from index date will be summarized by the K-M plot with the corresponding 95% CI.
  Index date is the date of the first dose of lorlatinib.
The real world intracranial progression free survival (rwICPFS) | 74 months from 1st April, 2018
  Time to real-world intracranial disease progression or death, whichever occurs first, during observation period from index date will be summarized by the K-M plot with the corresponding 95% CI.
  Index date is the date of the first dose of lorlatinib.

SECONDARY OUTCOMES:
Number and proportion of patients receiving each regimen of systemic anti-cancer therapy | 74 months from 1st April, 2018
  The percentage of patients with each systemic anticancer therapy for lung cancer.
Mean (SD), median (interquartile range, IQR), minimum and maximum value of duration of therapy (DoT) of lorlatinib | 74 months from 1st April, 2018
  Time to real-world discontinuation of lorlatinib or death, whichever occurs first, during observation period from index date will be summarized by the K-M plot with the corresponding 95% CI.
  Index date is the date of the first dose of lorlatinib.
Number and proportion of patients receiving concomitant antihyperlipidemic agents | 74 months from index date; index date is the date of the first dose of lorlatinib
  The number and percentage of patients receiving antihyperlipidemic agents received along with lorlatinib during the same treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Inc, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7461048